CLINICAL TRIAL: NCT05795023
Title: A Longitudinal Study to Evaluate the Correlation Between Oculometric Measures and MDS-UPDRS Over Time in a Cohort of Patients With Idiopathic Parkinson's Disease (PD)
Brief Title: A Longitudinal Evaluation of Oculometric Measures and Clinical Assessment Over Time in PD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLight (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL/PD/2022-3
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All patients will be assessed with MDS-UPDRS and oculometric examination over time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD patients (Experimental): Men and women with idiopathic PD (Hoehn & Yahr scale 1-3) aged 18-85 years
  Interventions: Other: NeuraLight

INTERVENTIONS:
Other: NeuraLight — NeuraLight software-based platform

SUMMARY:
This is a prospective study in a cohort of about 30 patients with Idiopathic Parkinson's disease, who will be evaluated with a clinical assessment and an oculometric examination during a time period with specific intervals.

This study aims to evaluate the correlation between oculometric measures and clinical assessment over time.

DETAILED DESCRIPTION:
This is an observational prospective cohort study, in a cohort of up to 30 patients with idiopathic PD. The aim of this study is to demonstrate that oculometric measures are able to detect patient deterioration faster than can be detected using the currently available clinical assessment tools. In addition, to evaluate the correlation between oculometric measures and Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score over time ,in subjects who meet the inclusion and exclusion criteria, and who provide a signed Informed Consent. All patients will be assessed using MDS-UPDRS over a period of 9 months (4 assessments, at 0, 3, 6, 9 months). During this time period, every subject who consents will undergo a NeuraLight session including oculometric measurements and eye-tracking recordings using a novel software-based platform and an eye- tracking system (Tobii, CE-marked class B approved device) (approx. 30 minutes). The oculometric evaluation will occur during the first 3 months for every patient every 2 weeks (+3 days), and then after 6 months and 9 months from enrollment (+3 days), (9 tests in total). All assessments will be performed during a clinic visit unless authorized to be conducted remotely. During the study, the sponsor will be blinded to the private details of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with idiopathic PD (Hoehn & Yahr scale 1-3)
* Age between 18 and 85 years old
* Normal or corrected vision
* Ability to follow instructions
* Willing and able to sign an informed consent form

Exclusion Criteria:

* Inability to sit for 30 minutes on a chair in a calm manner
* Personal or 1st degree relative history of epilepsy
* Additional neurological diseases
* Drug or alcohol abuse (except for using medical cannabis during 24 hours prior NL examination date)
* Pregnancy or a potential pregnancy (self-declaration)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change of saccadic latency over time as evaluated during visits | 12 months
  Difference between saccadic latency (ms) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Change of anti-saccadic error rates over time as evaluated during visits | 12 months
  Difference between anti-saccadic error rates (%) as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Change of smooth pursuit speed over time as evaluated during visits | 12 months
  Difference between smooth pursuit speed (ms)as quantified during each visit by the NeuraLight test measured using a statistical comparison of values (e.g. t-test, ANOVA), p>0.05) over time during study period
Correlation between MDS-UPDRS score and its parts with saccadic latency | 12 months
  The correlation between MDS-UPDRS score and its parts with saccadic latency (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at visits
Correlation between MDS-UPDRS score and its parts with anti-saccadic error rates | 12 months
  The correlation between MDS-UPDRS score and its parts with anti-saccadic error rates (%), measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at visits
Correlation between MDS-UPDRS score and its parts with smooth pursuit | 12 months
  The correlation between MDS-UPDRS score and its parts with smooth pursuit speed (ms) measured using R-Square (high correlation>0.5, moderate correlation 0.2-0.5, low correlation<0.2), p<0.05) according to the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at visits

SECONDARY OUTCOMES:
Using the retrieved data of collected NeuraLight oculometric measures for calibration of prediction models of MDS-UPDRS clinical endpoint | 12 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of MDS-UPDRS with a relative root mean square error (RMSE) of <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Gurevich, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Movement Disorders Unit, Sourasky Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No